CLINICAL TRIAL: NCT00271401
Title: A Multicenter, Randomized Trial Evaluating 30-day and 6-month Clinical Outcomes With Three Different Treatment Strategies (Coronary Angioplasty + Abciximab, Intracoronary Stent + Abciximab, and Intracoronary Stent + Placebo) in Patients Undergoing Percutaneous Coronary Intervention
Brief Title: A Study Comparing the Efficacy and Safety of Intracoronary Stenting With or Without Abciximab, an Anti-Platelet Therapy, and Conventional Coronary Angioplasty With Abciximab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006265
Record Dates: First submitted 2005-12-30; First posted 2006-01-02 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Angioplasty, Transluminal, Percutaneous Coronary
Keywords: Stents; Angioplasty, Transluminal, Percutaneous Coronary
MeSH Terms: interventions — Angioplasty; Heparin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Angioplasty With Abciximab Plus Low-Dose Heparin (Experimental): Participants will receive conventional angioplasty/atherectomy along with bolus abciximab 0.25 milligram per kilogram (mg/kg) of body weight followed by a 0.125 microgram per kilogram per minute (mcg/kg/minute) infusion for 12 hours plus 7 unit per kilogram per hour (U/kg/hr) continuous infusion of heparin.
  Interventions: Other: Angioplasty; Drug: Abxicimab; Drug: Heparin
- Intracoronary Stent With Reo Pro Plus Low Dose Heparin (Experimental): Participants will receive intracoronary stent along with receive bolus abciximab 0.25 mg/kg of body weight followed by a 0.125 mcg/kg/minute infusion for 12 hours plus 7 U/kg/hr continuous infusion of heparin (low dose).
  Interventions: Other: Intracoronary Stent; Drug: Abxicimab; Drug: Heparin
- Intracoronary Stent With Placebo Plus Standard Dose Heparin (Placebo Comparator): Participants will receive intracoronary stent along with bolus placebo followed by placebo infusion for 12 hours plus 10 U/kg/hr continuous infusion of heparin (standard dose).
  Interventions: Other: Intracoronary Stent; Drug: Heparin; Drug: Placebo

INTERVENTIONS:
Other: Angioplasty
  Arms: Angioplasty With Abciximab Plus Low-Dose Heparin
Other: Intracoronary Stent
  Arms: Intracoronary Stent With Placebo Plus Standard Dose Heparin; Intracoronary Stent With Reo Pro Plus Low Dose Heparin
Drug: Abxicimab
  Arms: Angioplasty With Abciximab Plus Low-Dose Heparin; Intracoronary Stent With Reo Pro Plus Low Dose Heparin
Drug: Heparin
Drug: Placebo
  Arms: Intracoronary Stent With Placebo Plus Standard Dose Heparin

SUMMARY:
The purpose of this study is to compare the effectiveness and safety of intracoronary stenting with or without abciximab, an anti-platelet therapy, and conventional coronary angioplasty with abciximab in patients undergoing percutaneous coronary intervention.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled study evaluating the safety and effectiveness of intracoronary stenting with or without abciximab, an anti-platelet therapy, and conventional coronary angioplasty with abciximab in patients undergoing percutaneous coronary intervention. Patients will be randomly assigned to one of three treatment groups: coronary angioplasty plus abciximab, intracoronary stent plus abciximab, or intracoronary stent plus placebo. The primary measures of effectiveness will be a 30-day composite, clinical outcome as determined by the number of deaths, myocardial infarctions, or urgent repeat revascularizations. Please see attached results.

Patients will receive one of three different treatments: Coronary angioplasty plus abciximab; Intracoronary stent plus abciximab; or Intracoronary stent plus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for elective or urgent percutaneous coronary intervention
* Who are suitable candidates for either conventional angioplasty or primary intracoronary stent implantation
* Having a target artery (native or graft) stenosis of >= 60% (visual estimation)

Exclusion Criteria:

* Patients with acute ST-segment elevation myocardial infarction within the previous 12 hours
* With a planned staged procedure or having an unprotected left main coronary artery stenosis > 50%
* With active internal bleeding, having a condition that may increase the risk of bleeding, or receiving ongoing treatment with an oral anticoagulant at the time of study entry
* Having had a percutaneous coronary intervention within the previous 3 months or prior intracoronary stent placement in a target vessel
* Having hypertension with systolic blood pressure > 180 mm Hg or diastolic blood pressure > 100 mm Hg at the time of study entry, or a platelet count < 100,000/μL at baseline

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2399 (Actual)
Dates: Start 1996-07; Primary Completion 1997-09 (Actual); Study Completion 1997-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants With any one of these: Deaths, Myocardial Infarctions, or Urgent Repeat Revascularizations | Up to 30 days

SECONDARY OUTCOMES:
Number of Particpants with Angiographic Outcome, Death or Myocardial Infraction and Cardiovascular Functional Status | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.

REFERENCES:
- [Result] Topol EJ, Mark DB, Lincoff AM, Cohen E, Burton J, Kleiman N, Talley D, Sapp S, Booth J, Cabot CF, Anderson KM, Califf RM. Outcomes at 1 year and economic implications of platelet glycoprotein IIb/IIIa blockade in patients undergoing coronary stenting: results from a multicentre randomised trial. EPISTENT Investigators. Evaluation of Platelet IIb/IIIa Inhibitor for Stenting. Lancet. 1999 Dec 11;354(9195):2019-24. doi: 10.1016/s0140-6736(99)10018-7. PMID 10636365
- [Result] EPISTENT Investigators. Randomised placebo-controlled and balloon-angioplasty-controlled trial to assess safety of coronary stenting with use of platelet glycoprotein-IIb/IIIa blockade. Lancet. 1998 Jul 11;352(9122):87-92. doi: 10.1016/s0140-6736(98)06113-3. PMID 9672272